CLINICAL TRIAL: NCT03424551
Title: Vibration-induced Reflex Responses and Estimation of Tonic Vibration Latency
Brief Title: Vibration Induced Reflex Responses and Estimation of TVR
Acronym: VIRR&TVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IstPMRTRH-BMR1
Record Dates: First submitted 2018-01-24; First posted 2018-02-07 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Muscle; Physiology
Keywords: vibration; muscle spindle; H reflex; tonic vibration reflex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vibrator (Experimental): Local or Whole body vibration was applied at six different frequencies to Healthy control and spastic spinal cord injury. For local vibration, vibration frequencies were 50, 85, 140, 185, 235 and 265 Hz . For whole body vibration, vibration frequencies were 35, 37, 39, 41, 43 and 45 Hz
  Interventions: Device: vibrator

INTERVENTIONS:
Device: vibrator — Local or whole body vibration was applied at six different frequencies
  Other Names: cyclic mechanical loading

SUMMARY:
The aim of this study is to estimate tonic vibration latency and whole body vibration reflex latency

DETAILED DESCRIPTION:
This study was included 17 patients with spastic spinal cord lesions and 23 healthy control.

Soleus T-reflex, soleus H-reflex, soleus tonic vibration reflex (TVR), and reflex muscle response induced by whole body vibration was evaluated this study. To obtain the H-reflex response, the tibial nerve in the popliteal region was stimulated by using a stimulator (FE155 Stimulator HC ADInstrument, Oxford UK) with 1 ms-pulse current. The records was taken with the Ag / AgCl electrodes (Kendall ®Coviden, self-adhesive electrodes) placed on skin according to the SENIAM protocol. To obtain T-reflex response, an electronic reflex hammer (Elcon 100-150 Germany) was used. After H-reflex and T reflex records at rest, to obtain Tonic vibration reflex, local vibration was applied to the Achilles tendon at 50, 85, 140, 185, 235 and 265 Hz. To obtain the reflex response induced by Whole body vibration, vibration was applied at 35, 37, 39, 41, 43 and 45 Hz. Tibial nerve stimulation was performed again to determine Hmax during whole body vibration and local vibration.H-reflex records was taken while the subject is sitting on a chair.

The data was recorded with the PowerLab data acquisition device (ADInstrument Oxford UK). For Whole-body vibration, PowerPlate Pro5 (London UK) was used.

ELIGIBILITY:
Inclusion Criteria spinal cord injury patients:

* Spastic spinal cord lesion
* Patients between the ages of 20 and 45

Exclusion Criteria for spinal cord injury patients

* Accompanying trauma

  1. Lower extremity fracture
  2. Lower extremity peripheral nerve lesions
  3. Head trauma
* Autonomic dysreflexia
* Heterotopic ossification
* Lesions in calf skin
* Excessive spasticity (Ashwort4) / Contracture (knee, hip, footbath)
* Peripheral nerve-vascular diseases / muscle diseases
* Pressure ulcer (> Grade 2)

Inclusion criteria for Control

* Ages 20 and 45 old years
* Both sex
* Healthy volunteers

Exclusion Criteria for Control

* Pregnant women

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Presynaptic inhibition level | 1 day
  Change in Hmax amplitude during vibration

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa A Yıldırım, MD, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ashby P, Verrier M, Lightfoot E. Segmental reflex pathways in spinal shock and spinal spasticity in man. J Neurol Neurosurg Psychiatry. 1974 Dec;37(12):1352-60. doi: 10.1136/jnnp.37.12.1352. PMID 4375172
- [Background] Alizadeh-Meghrazi M, Masani K, Zariffa J, Sayenko DG, Popovic MR, Craven BC. Effect of whole-body vibration on lower-limb EMG activity in subjects with and without spinal cord injury. J Spinal Cord Med. 2014 Sep;37(5):525-36. doi: 10.1179/2045772314Y.0000000242. Epub 2014 Jul 1. PMID 24986541
- [Background] Karacan I, Cidem M, Cidem M, Turker KS. Whole-body vibration induces distinct reflex patterns in human soleus muscle. J Electromyogr Kinesiol. 2017 Jun;34:93-101. doi: 10.1016/j.jelekin.2017.04.007. Epub 2017 Apr 24. PMID 28457998
- [Background] Karacan I, Cidem M, Yilmaz G, Sebik O, Cakar HI, Turker KS. Tendon reflex is suppressed during whole-body vibration. J Electromyogr Kinesiol. 2016 Oct;30:191-5. doi: 10.1016/j.jelekin.2016.07.008. Epub 2016 Jul 25. PMID 27485766
- [Background] Cakar HI, Cidem M, Sebik O, Yilmaz G, Karamehmetoglu SS, Kara S, Karacan I, Turker KS. Whole-body vibration-induced muscular reflex: Is it a stretch-induced reflex? J Phys Ther Sci. 2015 Jul;27(7):2279-84. doi: 10.1589/jpts.27.2279. Epub 2015 Jul 22. PMID 26310784
- [Background] Karamehmetoglu SS, Karacan I, Cidem M, Kucuk SH, Ekmekci H, Bahadir C. Effects of osteocytes on vibration-induced reflex muscle activity in postmenopausal women. Turk J Med Sci. 2014;44(4):630-8. PMID 25551934
- [Background] Cidem M, Karacan I, Diracoglu D, Yildiz A, Kucuk SH, Uludag M, Gun K, Ozkaya M, Karamehmetoglu SS. A Randomized Trial on the Effect of Bone Tissue on Vibration-induced Muscle Strength Gain and Vibration-induced Reflex Muscle Activity. Balkan Med J. 2014 Mar;31(1):11-22. doi: 10.5152/balkanmedj.2013.9482. Epub 2014 Mar 1. PMID 25207162
- [Background] Cakar HI, Cidem M, Kara S, Karacan I. Vibration paradox and H-reflex suppression: is H-reflex suppression results from distorting effect of vibration? J Musculoskelet Neuronal Interact. 2014 Sep;14(3):318-24. PMID 25198227